CLINICAL TRIAL: NCT04995861
Title: A Comparison Between The Analgesic Efficacy of Adductor Canal Block Alone and Adductor Canal With IPACK (Interspace Between Popliteal Artery and Capsule of the Knee) Block for Knee Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohammed Shabayek, Assistant lecturer of anesthesia , intensive care and pain management, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AinShamsU Shabayek MD
Record Dates: First submitted 2021-07-24; First posted 2021-08-09 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Nerve Blocks

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (adductor canal only) (Active Comparator): Will recieve adductor canal block only
  Interventions: Procedure: Adductor canal block and IPACK block
- Group AB (adductor canal + IPACK) (Active Comparator): Will recieve both adductor canal block and IPACK
  Interventions: Procedure: Adductor canal block and IPACK block

INTERVENTIONS:
Procedure: Adductor canal block and IPACK block — Peripheral nerve blocks

SUMMARY:
A comparison between The analgesic efficacy of adductor canal block alone and adductor canal with IPACK (interspace between popliteal artery and capsule of the knee) block for knee surgeries

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing knee surgery i.e. arthroscopy, total knee replacement, ACL repair.
* ASA physical status I to III
* Sex (males and females)
* Age 21-70 years.

Exclusion Criteria:

* Hypersensitivity to local anesthetics. Preexisting peripheral neuropathy. Infection near site of infections e.g. osteomyelitis, septic knee joint. Etc. Patient refusal. PAny contraindications for spinal anesthesia. ( eg: coagulopathy, use of anticoagulants

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-09-20 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of post operative pain | One year
  Using visual analogue scale (VAS) (scale 0-10, where 0 = no pain and 10 = worst imaginable pain)

SECONDARY OUTCOMES:
Range of movement and ambulation | One year
  the range of movement (ROM) by assessing the degree of knee extension one day after the surgery, and ambulation distance assessed by the number of steps walked by the patient three days after the surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided